CLINICAL TRIAL: NCT01027377
Title: An Open-Label, Crossover, Dose-Escalation, and Multi-Center Study to Determine the Safety, Tolerability, and Pharmacokinetic of a Single Intravenous Injection of rFVIIIFc in Previously Treated Patients With Severe Hemophilia A
Brief Title: Study of Recombinant Factor VIII Fc Fusion Protein (rFVIIIFc) in Subjects With Severe Hemophilia A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 998HA101
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-08

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Cohort to receive a single low dose intravenous injection of commercially available rFVIII with safety and PK assessments followed by a single low dose intravenous injection of rFVIIIFc with safety and PK assessments
  Interventions: Drug: rFVIIIFc
- B (Experimental): Cohort to receive a single high dose intravenous injection of commercially available rFVIII with safety and PK assessments followed by a single high dose intravenous injection of rFVIIIFc with safety and PK assessments
  Interventions: Drug: rFVIIIFc

INTERVENTIONS:
Drug: rFVIIIFc — Single dose
  Other Names: Recombinant Factor VIII fusion protein
  Arms: A
Drug: rFVIIIFc — Single dose
  Other Names: Recombinant Factor VIII fusion protein
  Arms: B

SUMMARY:
The study is to investigate the safety, tolerability, and pharmacokinetics (the determination of the concentration of the administered drug in blood over time) of recombinant Factor VIII Fc fusion protein (rFVIIIFc) in previously-treated subjects with severe hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

1. Male and 12 years of age and older and weigh at least 40 kg
2. Diagnosed with severe hemophilia A (baseline Factor VIII level less than 1%)
3. History of at least 100 exposure days to any Factor VIII product

Exclusion Criteria:

1. History of Factor VIII inhibitors
2. Kidney or liver dysfunction
3. Diagnosed with another coagulation defect other than hemophilia A

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by physical examination, vital signs, laboratory changes overtime, adverse events, and assessment of inhibitor (Bethesda) and antibody development against rFVIIIFc. | 78 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters will be measured such as, but not limited to Tmax, Cmax, t1/2, CL, Vd, AUC, MRT, and incremental recovery. | 78 weeks
To determine the pharmacokinetics parameters after single administration of 25 and 65 IU/kg of rFVIIFc compared to advate | 78 weeks
To determine the pharmacodynamic activity of FVIII over time for both doses of rFVIIIFc | 78 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Waltham, Massachusetts
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Seattle, Washington
- Research Site, Hong Kong, Hong Kong
- Research Site, Tel Aviv, Israel

REFERENCES:
- [Derived] Katragadda S, Neelakantan S, Diao L, Wong N. Population Pharmacokinetic Analysis of Recombinant Factor VIII Fc Fusion Protein in Subjects With Severe Hemophilia A: Expanded to Include Pediatric Subjects. J Clin Pharmacol. 2021 Jul;61(7):889-900. doi: 10.1002/jcph.1854. Epub 2021 Apr 14. PMID 33719084
- [Derived] Powell JS, Josephson NC, Quon D, Ragni MV, Cheng G, Li E, Jiang H, Li L, Dumont JA, Goyal J, Zhang X, Sommer J, McCue J, Barbetti M, Luk A, Pierce GF. Safety and prolonged activity of recombinant factor VIII Fc fusion protein in hemophilia A patients. Blood. 2012 Mar 29;119(13):3031-7. doi: 10.1182/blood-2011-09-382846. Epub 2012 Jan 5. PMID 22223821